CLINICAL TRIAL: NCT04892680
Title: Enhancing Cardiometabolic Care Study
Brief Title: Impact of a Digital Self-Management Program on A1C for Individuals With Type 2 Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated prematurely due to operational futility.
Sponsor: Omada Health, Inc. (Industry)
Collaborators: Sutter Health (Other); Palo Alto Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.082-1
Record Dates: First submitted 2021-05-04; First posted 2021-05-19 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; diabetes education; digital health; behavior modification
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Diabetes Self-Management Education and Support (DSMES) Program (Experimental): Participants will receive access to a 6-month online DSMES program that includes several components that are standard to DSMES. Participants receive online curriculum, access to a live Certified Diabetes Care and Education Specialist (CDCES), interactive group message forums, and connected devices for monitoring food intake, weight, physical activity and glucose levels.
  Interventions: Behavioral: Online Diabetes Self-Management Education and Support (DSMES) Program
- Matched Control (No Intervention): A de-identified dataset of control subjects matched on baseline demographics and clinical characteristics will be cultivated for comparison to the active intervention arm.

INTERVENTIONS:
Behavioral: Online Diabetes Self-Management Education and Support (DSMES) Program — Digital delivery of a DSMES program designed to build self-management skills and support diabetes management. Recipients have access to online curriculum, a live CDCES, group-based communication forums, and connected technology to track weight, food intake, physical activity and glucose levels.
  Arms: Online Diabetes Self-Management Education and Support (DSMES) Program

SUMMARY:
The goal of this study is to evaluate a digital chronic disease self-management program designed to provide virtual support and guidance for patients with type 2 diabetes.

DETAILED DESCRIPTION:
Approximately 45% of patients with type 2 diabetes do not achieve adequate glycemic control (A1C < 7%). When diabetes is uncontrolled, complications develop that threaten health and endanger life. This study will make an effort to address this growing health challenge and to reduce the burden of diabetes in this population. More broadly, this study will have important implications and benefits for the growing diabetes population in the U.S. Study results will inform future interventions to reduce diabetes and improve outcomes. A better understanding of the efficacy of a digital chronic disease self-management program will directly benefit the participants of the program but, in the future, has the potential to more broadly benefit this population throughout the nation.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age and less than 65 years of age
* Overweight (BMI ≥ 25 kg/m2, or BMI ≥ 23 kg/m2 if of Asian descent)
* Uncontrolled type 2 diabetes (HbA1C ≥7.5% and ≤12%)
* Diagnosed with type 2 diabetes at least 6 months ago, but not more than 10 years ago
* Has a compatible smartphone running either Android Operating System 5.0 or higher, or iPhone 7 or later, running iOS 11 or higher.
* Willing to set up an online account
* An email address in regular use
* Ambulatory (e.g., living at home and not in a skilled nursing facility)
* Able to speak, understand, and read English

Exclusion Criteria:

* A diagnosis of Type 1 diabetes
* Currently pregnant or postpartum (within 4 weeks)
* Currently using a continuous glucose monitor to manage diabetes
* Known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin
* Skin lesions, scarring, redness, infection or edema at the continuous glucose monitor application sites (upper arm) that could interfere with sensor placement or the accuracy of interstitial glucose measurements
* An active eating disorder such as anorexia or bulimia (not including binge-eating disorder) for which he/she has received treatment in the past 12 months
* Alcohol or substance abuse that impairs ability to participate in the program
* Unable to engage in physical activity for more than 2 months over the next 6 months (i.e. due to injury or recent or planned surgery)
* Any of the following in the past 3 months AND are not medically cleared by your physician to exercise: Transient ischemic attack or stroke; Heart attack (myocardial infarction); Hospitalization for congestive heart failure; Cardiac surgery (such as coronary artery bypass grafting (CABG), coronary artery stenting); Bariatric/gastric bypass surgery
* Received a solid Organ Transplant (kidney, liver, etc.) within the past 6 months
* Recent (within the last 6 months) or planned cancer treatment (chemotherapy, radiation, bone marrow transplant, cancer-related surgery - not including hormonal chemotherapy, such as tamoxifen).
* On dialysis treatment
* Taking steroids or prednisone (high doses) or getting cortisone injection
* Stage 4-5 Chronic Kidney Disease
* Class 3-4 Congestive Heart Failure
* Participation in diabetes education in the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c at 6 months from baseline | Baseline, 6 months
  Non-fasting venous blood sample

SECONDARY OUTCOMES:
Change in weight at 6 months from baseline | Baseline, 6 months
  Percentage of body weight loss
Change in medication adherence at 6 months from baseline | Baseline, 6 months
  The Adherence Estimator, a three-item self-report questionnaire, will be used to assess medication adherence

OTHER OUTCOMES:
Health care utilization at 6 and 12 months from baseline | Baseline, 6 months, 12 months
  Patient electronic health record data will be collected to examine the impact on short-term health care utilization

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Li, PhD, Principal Investigator — Palo Alto Medical Foundation
Locations (1):
- Palo Alto Medical Foundation Research Institute, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No